CLINICAL TRIAL: NCT05964465
Title: Mechanisms of Smell Improvement With Dupilumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Shaun Nguyen, Professor and Director of Clinical Research, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00125142
Record Dates: First submitted 2023-02-15; First posted 2023-07-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Chronic Rhinosinusitis; Nasal Polyps; dupilumab
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): The treatment group will receive dupilumab at 300mg SC Q2weeks. The first dose will be administered via subcutaneous injection in clinic at baseline. Subjects will self-administer study drug (dupilumab 300 mg) subcutaneous every 2 weeks after initial dosing at visit 2.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Monoclonal antibody blocking interleukin 4 and interleukin 13

SUMMARY:
This study seeks to explore the mechanism through which dupilumab improves olfactory cleft inflammation in patients with chronic sinusitis with nasal polyps (CRSwNP). The investigators expect this study to provide convincing evidence that dupilumab improves clinical olfaction via direct reduction in olfactory cleft inflammation.

DETAILED DESCRIPTION:
Post-marketed administration of dupilumab (FDA approved medication for CRSwNP) in patients with Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) will result in significant improvement in objective measures of olfactory cleft inflammation and psychophysical olfaction. The investigators seek to explore the mechanism through which dupilumab improves olfactory cleft inflammation in patients with CRSwNP. The investigators also want to determine whether change in olfactory cleft inflammation correlates with improvement in olfaction (one of the cardinal symptoms of CRSwNP) at 3 months. The investigators hypothesize that after 3 months of treatment with dupilumab, non-inflammatory factors will explain a significant degree of variation in residual clinical olfaction. Additionally, the investigators want to explore the determinants of ongoing olfactory loss after 3 months of treatment with attention to non-inflammatory factors. The investigators expect this study to provide convincing evidence that dupilumab improves clinical olfaction via direct reduction in olfactory cleft inflammation. Specifically, the investigators expect to show that reduction in olfactory cleft inflammation is the result of reduction in IL13 levels in olfactory cleft mucus. Finally, the investigators expect to show that most of the variation in post-treatment olfaction can be explained by non-inflammatory measures that are independent of CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Meet criteria for CRSwNP as defined by ICAR-21
* 2 out of 4 cardinal symptoms for ≥12 weeks
* Visible evidence of inflammation on endoscopy or imaging
* Bilateral visible nasal polyps ≥1 in each nasal cavity (0-4 scale each side)
* Olfaction score ≥1 (0-3 scale)
* Candidate for treatment with dupilumab for CRSwNP
* Elected to proceed with dupilumab for treatment of CRSwNP

Exclusion Criteria:

* Prior use of dupilumab
* Previous treatment with another biologic medication for CRSwNP or asthma within 6 months
* Any nasal or sinus surgery within the last 3 months
* Oral corticosteroid use within the last 1 month
* Current pregnancy, breast-feeding, or plan to become pregnant during next 3 months
* Presence of antrochoanal nasal polyps; acute rhinosinusitis; upper respiratory infection;
* Allergic granulomatous angiitis/eosinophilic granulomatosis with polyangiitis;
* Granulomatosis with polyangiitis; cystic fibrosis; Young syndrome;
* Kartagener syndrome; or dyskinetic cilia syndrome
* Poorly controlled asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in volumetric olfactory cleft opacification based on CT. | 3 months post-treatment
  Non-contrast sinus computed tomography (CT) scans will be obtained at baseline and 3 month follow-up to provide 1mm cuts that can be formatted in coronal, sagittal, and axial planes. Volumetric analysis of the OC will be performed utilizing equally spaced coronal CT images per our previously described protocols. Total volume of the segmented 3-D olfactory cleft space will be calculated, as well as the volume of air within that space. The percent opacification will be defined as [1-(total volume of air/total volume of olfactory cleft)] multiplied by 100. Sinus opacification will be quantified using the Lund-Mackay CT scale.
Change in olfactory cleft endoscopy score based on nasalendoscopy. | 3 months post-treatment
  Subjects will have sinonasal endoscopy at baseline and every follow up visit. This procedure allows visual inspection of the sinus mucosal lining and grading of polyps, including the olfactory cleft. Results for each side will be recorded separately and combined for a final Olfactory Cleft Endoscopy Scale (OCES) that ranges from 0-20, with higher scores representing increased disease severity.
Change in olfactory cleft mucus cytokine levels | 3 months post-treatment
  Under endoscopic guidance, a 1 × 2-cm Leukosorb filter paper (Pall Scientific, Port Washington, NY) strip will be placed into the olfactory cleft of each side, and kept in place for 3 minutes, as described in earlier studies. This will be done at baseline, 2 weeks, and 3 months. Olfactory cleft mucus inflammatory cytokine levels will be detected using commercially available LegendPlex Th2 Cytometric Bead Array (BioLegend, San Diego, CA) following the manufacturer's recommended protocol. This panel will include IL4, IL13, IL5 cytokines (among others). The assay will be carried out according to manufacturers' instructions and as previously described. The samples will be read on a Guava easyCyte 8HT flow cytometer (EMD Millipore) and analysis performed with LegendPlex software. Total IgE will be quantified via ELISA (GenWay Biotech. Inc, San Diego, CA).
Change in Lund-Kennedy endoscopy score. | 3 months post-treatment
  Subjects will have sinonasal endoscopy at baseline and every follow up visit. This procedure allows visual inspection of the sinus mucosal lining and grading of polyps, including the olfactory cleft. Results for each side will be recorded separately and combined for a final Lund-Kennedy endoscopy score (LKES) that ranges from 0-20, with higher scores representing increased disease severity.
Change in overall polyp score from sinonasal endoscopy | 3 months post-treatment.
  Overall polyp score on a 0-4 scale for each nostril (summed 0-8).

SECONDARY OUTCOMES:
Correlation between change in olfactory cleft mucus IL13 level and Sniffin Sticks TDI | 3 months post-treatment
  Quantitative psychophysical olfactory testing will be performed using the "Sniffin' Sticks" test (Burghardt, Wedel, Germany). Testing will be performed by trained clinical research coordinators who routinely perform objective olfactory testing and will be done in a blinded fashion. This commercially available test battery measures odor threshold (OT), odor discrimination (OD) and odor identification (OI). The results will be combined for an overall TDI score. TDI will be correlated with OC IL13 levels.
Correlation between change in IL13 level and QOD-NS score | 3 months post-treatment
  Olfactory-specific QOL will be assessed using the previously validated, short, modified version of the Questionnaire of Olfactory Disorders (QOD-NS) survey. This instrument was validated by Mattos and Soler and has been found to have criterion validity, internal consistency, and excellent reproducibility.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia, Charlottesville, Virginia